CLINICAL TRIAL: NCT00270504
Title: Prospective, Randomized, Controlled, Multicenter Trial of the Memokath® 044TW Thermo-Expandable Stent for Maintaining Urethral Patency in Patients After Dilation or Internal Urethrotomy of Recurrent Stricture of the Bulbar Urethra
Brief Title: Memokath® 044TW Stent for Treatment of Urethral Stricture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pnn Medical DK (Industry)
Responsible Party: Director of Clinical and Regulatory, Pnn Medical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-044TWUS
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2008-12

CONDITIONS: Urethral Stricture
Keywords: Memokath; Urethral stricture; urethral stent; Bulbar urethral stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Memokath stenting — Urethral Stenting

SUMMARY:
The purpose of this study is to evaluate if the placement of a temporary urethral stent for up to 12 months, following dilation or internal urethrotomy (cutting open), results in a higher rate of urethral patency during the first year of follow-up when compared to the control group that does not receive a stent.

DETAILED DESCRIPTION:
Patients with bulbar urethral stricture are 2:1 randomised for either urethral dilation or internal urethrotomy with (treatment group) or without (control group) subsequent stenting. All patients are followed for up to one year at 4-6 weeks, 3, 6, 9 and 12 months with visual assessment (urethroscopy) of urethral patency at the treated segment of the urethra. The stent is removed at one year. In case of premature stent removal the patient is also followed for up to one year unless further intervention is decided.

Control patients are offered the stent treatment option if the stricture recurs within the observation period but this group is separately analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Males > 21 years of age
2. Recurrent stricture of the bulbar urethra:

   1. < 50 mm in length on urethrography; and which
   2. has a segment unable to accommodate a 16Fr flexible cystoscope
3. Healthy tissue on both sides of stent
4. Urinary flow in the abnormal range of the Siroky nomogram.
5. Written informed consent obtained prior to participation in the study
6. Patients must be available for all follow-up visits.

Exclusion Criteria:

1. Strictures:

   1. outside the bulbous urethra
   2. associated with, or suspected to be, urethral carcinoma
   3. secondary to pelvic distraction injuries
2. Inability to enlarge the bulbar urethral stricture to > 26 Fr.
3. Presence of any other urologic implant
4. Presence of urethral diverticuli
5. History of hypospadias repair
6. Presence or prior history of balanitis xerotica obliterans.
7. Uncontrolled bleeding disorder
8. Active urinary tract infection
9. Any urological condition that would be likely to require additional urethral instrumentation during the period of the investigation, including, but not limited to, benign prostatic hypertrophy requiring treatment; use of alpha blockers; active prostate cancer; an unevaluated elevated prostate-specific antigen (PSA); bladder malignancy; or any recurrent urinary stone formation.
10. Serum creatinine > 2.0 mg/dl or evidence of progressive renal disease
11. Concurrent participation in another clinical investigation
12. Current illness that might confound the results of this investigation
13. Inability to participate in all of the necessary study activities
14. Inability or unwillingness to return for all required follow-up visits
15. Inability or unwillingness to sign the patient informed consent document

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2002-12; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Stent/control effectiveness - urethral patency | 1 year

SECONDARY OUTCOMES:
Peak urinary flow rate | Immediate
Re-intervention | Short term
Standard survey instruments (QOL, IPSS etc.) | 15 mos
Stent placement success | immediate
Stent removal success | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Jordan, MD, Principal Investigator — Sentara/Engineers and Doctors
Locations (7):
- United States (7):
  - Jack McAninch, San Francisco, California
  - Mississippi Urology, Jackson, Mississippi
  - Cleveland Clinic, Cleveland, Ohio
  - Bryn Mawr Urology, Bryn Mawr, Pennsylvania
  - University Urological Associates, Providence, Rhode Island
  - Devine-Tidewater Urology, Norfolk, Virginia
  - Harborview Medical Center, Seattle, Washington